CLINICAL TRIAL: NCT03623321
Title: A 52-Week Open-label Extension Study of Pimavanserin in Adult and Elderly Subjects With Neuropsychiatric Symptoms Related to Neurodegenerative Disease
Brief Title: Extension Study of Pimavanserin in Adult Subjects With Neuropsychiatric Symptoms Related to Neurodegenerative Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-047; 2017-004439-36 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Neuropsychiatric Symptoms Related to Neurodegenerative Disease
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - pimavanserin (Experimental): Pimavanserin 34 mg is provided as 2×17 mg tablets as single dose, once daily by mouth. Dose adjustments of pimavanserin down to 20 mg (provided as 2×10 mg tablets as a single dose, once daily by mouth) and up to 34 mg are permitted based on Investigator assessment of clinical response.
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — • Pimavanserin 34 mg is provided as 2×17 mg tablets as single dose, once daily by mouth. Dose adjustments of pimavanserin down to 20 mg (provided as 2×10 mg tablets as a single dose, once daily by mouth) and up to 34 mg are permitted based on Investigator assessment of clinical response.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of pimavanserin in adult and elderly subjects with neuropsychiatric symptoms related to neurodegenerative disease exposed to open-label pimavanserin for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject satisfied all entry criteria for the antecedent pimavanserin study
2. Subject completed the antecedent study; or was participating in a pimavanserin study that the Sponsor ended early
3. Has a designated study partner/caregiver who meets the following requirements:

   1. In the Investigator's opinion, is in contact with the subject frequently enough to accurately report on the subject's symptoms and whether or not the subject is taking the study drug
   2. In the Investigator's opinion, is considered reliable in providing support to the subject to help ensure compliance with study treatment, study visits, and protocol procedures
   3. Is fluent in the local language in which study assessments will be administered
   4. Agrees to participate in study assessments, has the capacity to provide informed consent, and provides written consent to participate in the study
4. Subject is willing and able to provide informed consent.
5. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential (defined as either surgically sterilized or at least 1 year postmenopausal) or must agree to use a clinically acceptable method of contraception or be abstinent during the study and 1 month following completion of the study.

Exclusion Criteria:

1. Subject is judged by the Investigator or the Medical Monitor to be inappropriate for the study, due to AEs, medical condition, or noncompliance with investigational product or study procedures in the antecedent study, or is judged to be a danger to self or others
2. Is in hospice, is receiving end-of-life palliative care, or has become bedridden
3. Has any of the following ECG results at the EOT/ET visit of the antecedent study:

   a. If the subject is not on citalopram, escitalopram, or venlafaxine:

   i. QTcF >450 ms, if QRS duration <120 ms

   ii. QTcF >470 ms, if QRS duration ≥120 ms

   b. If the subject is on citalopram, escitalopram, or venlafaxine:

   i. QTcF >425 ms, if QRS duration <120 ms

   ii. QTcF >450 ms, if QRS duration ≥120 ms
4. Has a heart rate <50 beats per minute. If bradycardia is secondary to iatrogenic or treatable causes and these causes are treated, a heart rate assessment can be repeated at the EOT/ET visit of the antecedent study.
5. Has clinically significant laboratory abnormalities in the antecedent study that, in the judgment of the Investigator or Medical Monitor, would either:

   1. jeopardize the safe participation of the subject in the study; OR
   2. would interfere with the conduct or interpretation of safety or efficacy evaluations in the study
6. Is suicidal at Visit 1 (Baseline)
7. Has developed a medical condition that in the judgment of the Investigator, would increase the risk associated with taking study medication or significantly interfere with the conduct or interpretation of the study
8. Requires treatment with a medication or other substance that is prohibited by the protocol
9. Has a significant sensitivity or allergic reaction to pimavanserin or its excipients
10. Is an employee of ACADIA, or has a family member who is an employee of ACADIA

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (88):
- United States (17):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Syrentis Clinical Research, Santa Ana, California
  - Indago Research & Health Center Inc, Hialeah, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Global Medical Institutes, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - MediClear Medical & Research Center, Inc., Miami, Florida
  - Novel Clinical Research LLC, Miami, Florida
  - Laszlo J Mate, MD, PA, North Palm Beach, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - UNC Hospital, Chapel Hill, North Carolina
  - Insight Clinical Trials LLC, Shaker Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Central for Biomedical Research, LLC, Knoxville, Tennessee
- Bulgaria (6):
  - Centre for Mental Health Prof. Dr. Ivan Temkov, Lazur Compl., Park Ezero, Burgas
  - UMHAT Psych clin for gen psychiatry and addictions, Pleven
  - DCC Sv. Vrach and Sv. Sv. Kozma and Damyan, Sofia
  - Diagnostic Consultative Centre, 2, N. Vaptzarov Street, Varna
  - Diagnostic Consultative Centre-Mladost-Psychiatry, 15, Republika Blvd., Varna
  - Mental Health Center Vratza EOOD, 1 Belasitsa St., Vratsa
- Colombia (4):
  - E.S.E. Hospital Mental de Antioquia, Bello, Antioquia
  - Centr Investigaciones y Proyectos en Neurociencias, Barranquilla, Atlántico
  - Psynapsis Salud Mental S.A., Pereira, Risaralda Department
  - Centro de Investigaciones del Sistema Nervioso, Bogotá
- Czechia (5):
  - BRAIN-SOULTHERAPY s.r.o., Lekarna Jalta, Namesti Jana Masaryka 3113, Kladno
  - A-shine s.r.o./ Lekarna Centrum, Pilsen
  - AD71, s.r.o./Hostivarska lekarna, Prague
  - Axon Clinical, Prague
  - Neuropsychiatrie, s.r.o., Lekarna 6ka, Fajtlova 1, Prague
- Georgia (5):
  - Petre Sarajishvili Institute of Neurology LLC, Tbilisi
  - Pineo Medical Ecosystem LTD, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - Health Institute LLC, Tbilisi
  - S. Khechinashvili University Hospital LLC, Tbilisi
- Mexico (3):
  - Hospital Universitario Saltillo, Saltillo, Coahuila
  - Clinicos y Especialidades Medicas, Monterrey, Nuevo León
  - Christus Muguerza Hospital Sur, Monterrey, Nuevo León
- Poland (10):
  - MlynowaMed Sp Psych Dr. Joanna Lazarczyk, Bialystok
  - Wlokienniecza Med Sp Prak Lekarska Dromasz Markowski, Bialystok
  - Przychodnia Srodmiescie Sp. z.o.o., Bydgoszcz
  - ISPL Wieslaw Jerzy Cubala, Gdansk
  - NZOZ Syntonia Poradnia Zdrowia Psychicznego, ul. Cyprysowa 2F/ 9,10, Pruszcz, Gdansk
  - Krakowska Ak Neuro Sp.- Centrum Neuro Klinicznej, ul. Arianska 7/3, Krakow
  - Centrum Medyczne HCP Sp. zo.o, Poznan
  - Neuro-Care Sp. zo.o. sp. Komandytowa, Siemianowice Śląskie
  - Neuro-care, Siemianowice Śląskie
  - RCMed Oddzial Sochaczew, ul. _eromskiego 41A, Sochaczew
- Romania (3):
  - Spitalul clinic CF Constanta, Sectia Neurologie, Constanța
  - Med Anima SRL, Clinica de psihiatrie, Iași
  - S.C. Carpe Diem SRL, Sibiu
- Russia (11):
  - Regional Specialized Psychiatric Hospital #2, Tonnel’nyy, Kochubeev District
  - Federal Siberian Sci Clinical Center of Med and Bio, Krasnoyarsk
  - Mental Health Research Center, Moscow
  - City Clinical Hospital #34, Novosibirsk
  - Leningrad Regional Psychoneurological Dispensary, Roshchino
  - St. Nicholas the Wonder Worker Psychiatric Hospital, Saint Petersburg
  - FSBI NMRC PN n.a. V.M. Bekhterev, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Saratov City Clinical Hospital V. I. Razumovsky, Saratov
  - Stavropol Regional Clin Spec Psych Hospital #1, Stavropol
  - Clinic "Hundred Years", Tomsk
- Serbia (11):
  - CHC Dr Dragisa Misovic- Dedinje, Belgrade
  - Clinical Center of Serbia, Clinic for Psychiatry, Belgrade
  - Clinical Center of Serbia,Clinic for Neurology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinic for Psychiatric Diseases Dr. Laza Lazarevic, Belgrade
  - Klinicki Centar Srbije (KCS)- Klinika za nerurologiju, Belgrade
  - Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - Clinical Center Kragujevac, Clinic for Neurology, Kragujevac
  - Clinical Center Kragujevac,Clinic of Psychiatry, Kragujevac
  - Clinical Center Nis, Clinic for Psychiatry, Toponica
  - General Hospital Valjevo, Department for Neurology, Valjevo
- South Africa (2):
  - Neurology Practice, Pretoria, Gauteng
  - Flexivest Fourteen Research Centre Potocnik F C V, Durban, Western Cape
- Ukraine (11):
  - Dnipropetrovsk Regional Rehabilitation Hospital, Dnipro
  - Dnir. Regional Clinical Hospital n.a. Mechnikov, Dnipro
  - Ivano-Frankivsk Nat Med Uni Dep Psychiatry, Regional Hospital, Ivano-Frankivsk
  - Institute of Neruology, Nat Acad of Med Sci of UKR, Kharkiv
  - Institute of Neurology, Kharkiv
  - Municipal Non-Commercial Institution of Kharkiv Regional Council "Kharkiv Regional Clinical Psychiatric Hospital # 3" 46, Ac. Pavlova str., Kharkiv
  - Kyiv Regional Medical Incorp. Psychiatria, Center, Kyiv
  - Kyiv Regional Psychiatric and Narcological Medical Association 8, Vokzalna str., Glevakha, Kyiv
  - Ternopil Regional Communal Clinical Psychoneurological Hospital 14, Troleibusna str., Ternopil
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Male Department #7, Female Department #10, Vinnytsya National Medical University n.a. M.I.Pyrogov, Department of Psychiatry, Narcology and Psychotherapeutics, Vinnytsia
  - Municipal Unst Zaporizhzhya Reg Clinical Hosp Neurology, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension study to evaluate the long-term safety and tolerability of pimavanserin in patients with neuropsychiatric symptoms related to neurodegenerative disease, who had completed an antecedent study (ACP-103-046) or had participated in a pimavanserin study that the sponsor terminated early.
Groups:
- Pimavanserin: Pimavanserin 34 mg once daily (QD). Dose reductions to pimavanserin 20 mg and subsequent dose increases to 34 mg were allowed at any time, based on investigator assessment of clinical response of the patient.
Period: Overall Study
Arm/Group | Pimavanserin
Started | 595 (A total of 595 were enrolled in the study and started study treatment (pimavanserin).)
Completed | 452
Not Completed | 143
Not completed — Adverse Event | 32
Not completed — Death | 9
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 6
Not completed — Noncompliance with study drug | 6
Not completed — Use of prohibited medication | 3
Not completed — Physician Decision | 5
Not completed — Protocol Violation | 1
Not completed — Consent withdrawn by patient or legally accepted representative | 29
Not completed — Not further specified | 43

BASELINE CHARACTERISTICS:
Population: All patients enrolled and treated
Arm/Group | Pimavanserin
Number analyzed (Participants) | 595
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 348
  Male | 247
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 561
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  Colombia | 16
  Romania | 3
  United States | 197
  Czechia | 30
  Ukraine | 81
  Poland | 90
  Mexico | 9
  South Africa | 11
  Georgia | 25
  Bulgaria | 29
  Serbia | 36
  Russia | 68
Mini Mental State Examination total score [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a 30-item questionnaire to assess cognitive impairment. It focuses on areas of time and place of testing, repeating lists of words, arithmetic, language use and comprehension, and copying or drawing. Each of the 30 items has 2 possible values i.e. 0 (incorrect) or 1 (correct). The MMSE total score is derived as the sum of the item scores; it has a potential range of 0 to 30, with lower scores indicating greater cognitive impairment.
  units on a scale | 20.0 (5.16)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Number (%) of patients experiencing at least one TEAE
Time Frame: Treatment period and Follow-up period: 56 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin
Number analyzed (Participants) | 595
Participants | 238

ADVERSE EVENTS:
Time Frame: Treatment period and Follow-up period: 56 weeks
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 11/595
Serious Adverse Events (participants affected / at risk) | 37/595
Other Adverse Events (participants affected / at risk) | 0/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=595)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pneumonia necrotising (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Brain oedema (Nervous system disorders) | 2 (2)
Coma (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Aggression (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (2)
Disorientation (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03623321/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03623321/SAP_001.pdf